CLINICAL TRIAL: NCT01878344
Title: Effects of N-acetyl Cysteine on Major Cardiac and Cerebral Events in Patients Undergoing Primary Percutaneous Coronary Intervention Who Have Moderate to High Risk For Contrast Induced Nephropathy
Brief Title: Effects of N-acetyl Cysteine During Primary Percutaneous Coronary Intervention
Acronym: EASE-PRM-PCI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Ozaydin, MD, MD, Professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ozaydin290
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- n-acetyl cysteine (Experimental): 30 mg/kg/15 min intravenous bolus preprocedural and 50 mg/kg/8 h intravenous infusion during and after the procedure
  Interventions: Drug: NAC
- Saline (Placebo Comparator): 30 mg/kg/15 min intravenous bolus preprocedural and 50 mg/kg/8 h intravenous infusion during and after the procedure
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: NAC
  Arms: n-acetyl cysteine
Drug: Saline
  Arms: Saline

SUMMARY:
The aim of this study is to evaluate the effects of N-acetyl cysteine on major cardiac and cerebral events in patients undergoing primary percutaneous coronary intervention who have moderate to high risk for contrast induced nephropathy.

In a sub-group of patients coronary flow reserve will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute ST Elevation Myocardial Infarction undergoing Primary Percutaneous Coronary intervention Who Have Moderate to High Risk For Contrast Induced Nephropathy (Mehran Score ≥5)

Exclusion Criteria:

* Patients >18 years old with moderate to high risk for contrast induced nephropathy undergoing percutaneous coronary intervention
* Low risk for contrast induced nephropathy (Mehran Score <5)
* Use of nephrotoxic agents (NSAIDs, aminoglycosides,recent contrast injection...)
* Infection
* Pregnancy, Lactation
* Renal failure requiring dialysis
* Hepatic failure
* Allergy to NAC
* History of Asthma
* Chronic nitrate usage
* Malignancy
* Use of corticosteroids
* Leucocytosis,Thrombocytosis,Anemia
* Blood pressure of >180/100mmHg despite anti-hypertensive therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major cardiac and cerebral events | 1 year

SECONDARY OUTCOMES:
NAC side effects (Asthma exacerbation, Pruritus, Dyspnea) | during hospitalization at 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Mediterranean Region, Turkey (Türkiye)